CLINICAL TRIAL: NCT04543617
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study of Atezolizumab With or Without Tiragolumab (Anti-TIGIT Antibody) in Patients With Unresectable Esophageal Squamous Cell Carcinoma Whose Cancers Have Not Progressed Following Definitive Concurrent Chemoradiotherapy
Brief Title: A Study of Atezolizumab With or Without Tiragolumab in Participants With Unresectable Esophageal Squamous Cell Carcinoma Whose Cancers Have Not Progressed Following Definitive Concurrent Chemoradiotherapy
Acronym: SKYSCRAPER-07
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YO42137; 2020-001178-31 (EudraCT Number)
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Tiragolumab; atezolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Tiragolumab + Atezolizumab (Experimental): Participants will receive atezolizumab followed by tiragolumab.
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab
- Arm B: Tiragolumab Placebo + Atezolizumab (Experimental): Participants will receive atezolizumab followed by tiragolumab matching placebo.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab Matching Placebo
- Arm C: Tiragolumab Placebo + Atezolizumab Placebo (Placebo Comparator): Participants will receive matching placebos to tiragolumab and atezolizumab.
  Interventions: Drug: Tiragolumab Matching Placebo; Drug: Atezolizumab Matching Placebo

INTERVENTIONS:
Drug: Tiragolumab — Tiragolumab at a fixed dose of 600 milligrams (mg) administered by intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  Other Names: MTIG7192A, RO7092284
  Arms: Arm A: Tiragolumab + Atezolizumab
Drug: Atezolizumab — Atezolizumab at a fixed dose of 1200 mg administered by IV infusion Q3W on Day 1 of each 21-day cycle.
  Other Names: Tecentriq, RO5541267
  Arms: Arm A: Tiragolumab + Atezolizumab; Arm B: Tiragolumab Placebo + Atezolizumab
Drug: Tiragolumab Matching Placebo — Tiragolumab matching placebo administered by IV infusion Q3W on Day 1 of each 21-day cycle.
  Arms: Arm B: Tiragolumab Placebo + Atezolizumab; Arm C: Tiragolumab Placebo + Atezolizumab Placebo
Drug: Atezolizumab Matching Placebo — Atezolizumab matching placebo administered by IV infusion Q3W on Day 1 of each 21-day cycle.
  Arms: Arm C: Tiragolumab Placebo + Atezolizumab Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of tiragolumab plus atezolizumab compared with placebo in participants with unresectable esophageal squamous cell carcinoma (or those who are unable or unwilling to undergo surgery) and whose cancers have not progressed following definitive concurrent chemoradiotherapy (dCRT). Participants will be randomized in a 1:1:1 ratio to receive either tiragolumab plus atezolizumab (Arm A), tiragolumab matching placebo plus atezolizumab (Arm B), or double placebo (Arm C).

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Histologically or cytologically confirmed diagnosis of squamous cell carcinoma of the esophagus
* Unresectable disease ineligible for curative surgery based on the documented opinion of the qualified medical, surgical or radiation oncologist prior to dCRT and is not expected to undergo tumor resection during the course of the study
* dCRT treatment according to regional oncology guidelines for esophageal cancer
* Representative archival formalin-fixed, paraffin-embedded (FFPE) tumor specimens collected prior to initiation of dCRT
* Adequate hematologic and end-organ function prior to randomization
* Women of childbearing potential must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period, for 5 months after the final dose of atezolizumab/placebo, and for 90 days after the final dose of tiragolumab/placebo, whichever is later
* Men must agree to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agree to refrain from donating sperm during the treatment period and for 90 days after the final dose of tiragolumab/placebo.

Key Exclusion Criteria:

* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, anti-PD-L1 and anti-TIGIT therapeutic antibodies
* Any unresolved toxicity of National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥ 2 from the prior chemoradiation therapy with the exception of irreversible and manageable hearing loss
* Prior allogeneic stem cell or solid organ transplantation
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis
* Malignancies other than esophageal cancer within 2 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Treatment with any other investigational agent, including epidermal growth factor receptor (EGFR) inhibitors, with therapeutic intent for esophageal cancer prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Arm A vs Arm C: Investigator-Assessed Progression-Free Survival (PFS) | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 6 years)
Arm A vs Arm C: Overall Survival (OS) | From randomization to death from any cause (up to approximately 6 years)
Arm B vs Arm C: OS | From randomization to death from any cause (up to approximately 6 years)

SECONDARY OUTCOMES:
Arm B vs Arm C: Investigator-Assessed PFS | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 6 years)
Arm A vs Arm B: Investigator-Assessed PFS | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 6 years)
Arm A vs Arm B: OS | From randomization to death from any cause (up to approximately 6 years)
Independent Review Facility (IRF)-Assessed PFS | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 6 years)
Investigator-Assessed Confirmed Objective Response Rate (ORR) | From randomization up to approximately 6 years
IRF-Assessed Confirmed ORR | From randomization up to approximately 6 years
Investigator-Assessed Duration of Objective Response (DOR) | From the first occurrence of a documented confirmed objective response to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 6 years)
IRF-Assessed DOR | From the first occurrence of a documented confirmed objective response to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 6 years)
Percentage of Participants With Clinically Meaningful Changes in Physical Functioning, Role Functioning, Quality of Life (QoL) as Measured by EORTC QLQ-C30 | Up to approximately 6 years
  Clinically meaningful changes in physical functioning, role functioning, global health status (GHS)/QoL as measured by the European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30). EORTC QLQ-C30 is a self-reported measure, consisting of 30 questions that assess 5 aspects of participants functioning (physical, emotional, role, cognitive and social), 3 symptom scales (fatigue, nausea and vomiting, and pain), GHS and QoL, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties) within the previous week. Functioning and symptoms items are scored on a 4-point scale: 1=Not at all, 2=A little, 3=Quite a bit, 4=Very much. GHS and QoL items are scored on a 7-point scale: 1=Very poor, 2, 3, 4, 5, 6, 7=Excellent. Scores will be linearly transformed to a range of 0 to 100, with higher scores (i.e. closer to 100) reflecting better functioning, better GHS/QoL, and worse symptoms.
Percentage of Participants With Clinically Meaningful Changes in Dysphagia as Measured by EORTC QLQ-OES18 | Up to approximately 6 years
  Clinically meaningful changes in dysphagia as measured by the EORTC Quality of Life-Esophageal Cancer, Module 18 Questionnaire (EORTC QLQ-OES18). EORTC QLQ-OES18 is a modular supplement to the EORTC QLQ-C30 questionnaire for use in participants with esophageal cancer. EORTC QLQ-OES18 consists of 4 multiple-item scale (dysphagia, eating, reflux, and pain) and 6 single items (trouble swallowing saliva, choked when swallowing, dry mouth, trouble with taste, trouble with coughing, and trouble talking) with a recall period of the previous week. Each symptom item is scored on a 4-point scale: 1=Not at all, 2=A little, 3=Quite a bit, 4=Very much. Scores will be linearly transformed to a range of 0 to 100, with higher transformed scores (i.e. closer to 100) reflecting worse symptoms.
Percentage of Participants With Adverse Events (AEs) | Up to approximately 6 years
Serum Concentration of Tiragolumab | Predose and postdose on Day 1 of Cycle 1 (each cycle=21 days) and predose on Day 1 of Cycles 2, 3, 4, 8, 12 and 16 and at treatment discontinuation (TD) visit (up to approximately 6 years)
Serum Concentration of Atezolizumab | Predose and postdose on Day 1 of Cycle 1 (each cycle=21 days) and predose on Day 1 of Cycles 2, 3, 4, 8, 12 and 16 and at TD visit (up to approximately 6 years)
Percentage of Participants With Anti-drug Antibodies (ADAs) to Tiragolumab | Predose on Day 1 of Cycles (each cycle=21 days) 1, 2, 3, 4, 8, 12 and 16 and at TD visit (up to approximately 6 years)
Percentage of Participants With ADAs to Atezolizumab | Predose on Day 1 of Cycles (each cycle=21 days) 1, 2, 3, 4, 8, 12 and 16 and at TD visit (up to approximately 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial, Study Director — Hoffmann-La Roche
Locations (165):
- United States (3):
  - Florida Cancer Specialists - Fort Myers (Broadway), Fort Myers, Florida
  - Cancer Center of Kansas, Wichita, Kansas
  - Great Lakes Cancer Center, Williamsville, New York
- Argentina (3):
  - Instituto de Investigaciones Metabolicas (Idim), Buenos Aires
  - Fundacion Favaloro, Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), La Rioja
- Australia (3):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Austin Health, Heidelberg, Victoria
  - St John of God Hospital, Subiaco, Western Australia
- Austria (4):
  - Tiroler Landeskrankenanstalten Ges.M.B.H., Innsbruck
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Ordensklinikum Linz Barmherzige Schwestern, Linz
  - AKH - Medizinische Universität Wien, Vienna
- Belgium (3):
  - UZ Antwerpen, Edegem
  - UZ Leuven Gasthuisberg, Leuven
  - CHU de Liège (Sart Tilman), Liège
- China (35):
  - Anyang Tumor Hosptial, Anyang
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - Affiliated Hospital of Bengbu Medical College, Bengbu
  - Hunan Cancer Hospital, Changsha
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi
  - Changzhou Cancer hospital, Changzhou
  - Sichuan Provincial Cancer Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - Chongqing Sanxia Central Hospital, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Jieyang People's Hospital, Jieyang
  - Shandong Cancer Hospital, Jinan
  - Affiliated Hospital of Jining Medical University, Jining
  - The First People's Hospital of Lian Yun Gang, Lianyungang
  - Lishui Central Hospital, Lishui
  - The First Affiliated Hospital to Henan University of Science and Technology, Luoyang
  - Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - Liaoning cancer Hospital & Institute, Shenyang
  - Cancer Hospital Chinese Academy of Medical Sciences Shenzhen Center, Shenzhen
  - Hebei Medical University Fourth Hospital, Shijiazhuang
  - Tianjin Cancer Hospital, Tianjin
  - Wuhan Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Zhongshan Hospital Xiamen University, Xiamen
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - Subei People's Hospital of Jiangsu province, Yangzhou
- France (10):
  - CHRU De Brest - Hopital Morvan - Institut De Cancerologie Et D'Hematologie, Brest
  - CHU Dijon Bourgogne Hôpital François Mitterand, Dijon
  - Hopital Claude Huriez, Lille
  - Centre Leon Berard, Lyon
  - Hopital Timone Adultes, Marseille
  - Centre Antoine Lacassagne, Nice
  - European Hospital Georges Pompidou (HEGP), Paris
  - Hopital Du Haut-Leveque, Pessac
  - Chu La Miletrie, Poitiers
  - Hopital Rangueil, Toulouse
- Germany (7):
  - Universitätsklinikum Essen Klinik f.Strahlentherapie, Essen
  - Kliniken Essen-Mitte, Evang. Huyssens-Stiftung, Klinik für Internistische Onkologie / Haematologie, Essen
  - Klinik für Gastroenterologie und Gastrointestinale Onkologie der UMG, Göttingen
  - Universitaetsklinikum Leipzig, Leipzig
  - Med. Fak. d. Otto-von-Guericke-Universität, Magdeburg
  - Klinikum der Philipps-Universität Marburg, Marburg
  - Universitätsklinikum Klinik u.Poliklinik f.Strahlentherapie, Regensburg
- Greece (3):
  - Evgenidio Hospital "Agia Trias", Athens
  - Univ General Hosp Heraklion, Heraklion
  - Euromedical General Clinic of Thessaloniki, Thessaloniki
- Hungary (2):
  - Pécsi Tudományegyetem, Pécs
  - Szegedi Tudományegyetem, Szeged
- Israel (3):
  - Hadassah Ein Karem Hospital, Jerusalem
  - Rambam Health Corporation, Rambam
  - Tel Aviv Sourasky Medical Ctr, Tel Aviv
- Italy (4):
  - Università degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Ospedale Degli Infermi - Faenza, Faenza, Emilia-Romagna
  - Asu Fc S. M. Della Misericordia, Udine, Friuli Venezia Giulia
  - Istituto Oncologico Veneto IRCCS, Padua, Veneto
- Japan (15):
  - Aichi Cancer Center Hospital, Aichi
  - National Cancer Center Hospital East, Chiba
  - Hiroshima University Hospital, Hiroshima
  - Kobe University Hospital, Hyōgo
  - Yokohama City University Medical Center, Kanagawa
  - Kanagawa Cancer Center, Kanagawa
  - Tohoku University Hospital, Miyagi
  - Niigata Cancer Center Hospital, Niigata
  - Osaka International Cancer Institute, Osaka
  - The University of Osaka Hospital, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Keio University Hospital, Tokyo
- Kenya (2):
  - International Cancer Institute (ICI), Eldoret
  - The Aga Khan University-Kenya., Nairobi
- Morocco (3):
  - Centre Hospitalier Universitaire Hassan II, Fes
  - Centre Hospitalier Universitaire Mohamed VI, Marrakesh
  - Institut National D'oncologie Sidi Med Benabdellah, Rabat
- Tauranga Hospital, Clinical Trials Unit, Tauranga, New Zealand
- Poland (6):
  - Centrum Onkologii, Bydgoszcz
  - Centrum Onkologii Ziemi Lubelskiej Im. ?W. Jana Z Dukli, Lublin
  - Szpital Kliniczny MSWiA z Warmi?sko-Mazurskim Centrum Onkologii, Olsztyn
  - Wielkopolskie Centrum Onkologii im. Marii Sk?odowskiej-Curie, Późna
  - NIO im Marii Sklodowskiej-Curie, Warsaw
  - Dolno?l?skie Centrum Onkologii, Wroc?aw
- Portugal (3):
  - HUC, Coimbra
  - Centro Hospitalar do Porto ? Hospital de Santo António, Porto
  - IPO do Porto, Porto
- Russia (6):
  - Krasnoyarsk Regional Oncology Dispensary n.a. Krizhanovsky, Krasnoyarsk, Krasnodarskiy Kray
  - Russian Oncology Research Center n.a. N.N. Blokhin Dpt of Clinical Pharmacology and Chemotherapy, Moscow, Moscow Oblast
  - Republican Clinical Oncology Dispensary of Ministry of Healthcare of Tatarstan Republic, Kazan', Tatarstan Republic
  - City Oncological Hospital, Izhevsk, Udmurtiya Republic
  - Limited Liability Company "RC Medical", Novosibirsk
  - Regional Oncology Dispensary, Tomsk
- South Africa (3):
  - Limpopo Cancer Research Institute, Polokwane
  - Cancercare, Port Elizabeth
  - Eugene Marais Hospital, Pretoria
- South Korea (7):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Ajou University Medical Center, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (9):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña, LA Coruna
  - Hospital Univ. Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital La Fe, Valencia
- Switzerland (2):
  - Inselspital Bern, Insel-Gruppe AG, Bern
  - UniversitätsSpital Zürich, Zurich
- Taiwan (6):
  - Chang Gung Medical Foundation - Kaohsiung;Oncology, Kaohisung
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi-Mei Medical Centre, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (5):
  - Vajira Hospital, Bangkok
  - Chulalongkorn Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (6):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital, Adana
  - Ankara University Faculty of Medicine Cebeci Hospital, Ankara
  - Ankara City Hospital, Ankara
  - Ataturk University Medical Faculty Yakutiye Research Hospital Medical Oncology Department, Erzurum
  - Inonu University Faculty of Medicine Turgut Ozal Medical Center, Malatya
  - Van Yuzuncu Yil University Hospital, Van
- Ukraine (4):
  - Municipal Noncommercial Institution Regional Center of Oncology, Kharkiv, Kharkiv Governorate
  - Zhytomyr Regional Oncology Center, Zhytomyr, KIEV Governorate
  - Vinnytsya Regional Clinical Oncology Dispensary, Vinnytsia, Podolia Governorate
  - RCI Sumy Regional Clinical Oncological Dispensary, Sumy
- United Kingdom (7):
  - Royal Bournemouth Hospital, Bournemouth
  - Addenbrookes Hospital, Cambridge
  - Ninewells Hospital, London
  - Royal Marsden Hospital - Fulham, London
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Royal Marsden Hospital (Sutton), Sutton
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing